CLINICAL TRIAL: NCT00004771
Title: Phase II Study of Leuprolide and Testosterone for Men With Kennedy's Disease or Other Motor Neuron Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Ohio State University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11792; OSU-92H0325
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Spinal Muscular Atrophy; Amyotrophic Lateral Sclerosis; Spinobulbar Muscular Atrophy
Keywords: amyotrophic lateral sclerosis; motor neuron disease; neurologic and psychiatric disorders; rare disease; spinal and bulbar muscular atrophy; spinal muscular atrophy; Kennedy's Syndrome
MeSH Terms: conditions — Muscular Atrophy, Spinal; Amyotrophic Lateral Sclerosis; Bulbo-Spinal Atrophy, X-Linked; Motor Neuron Disease; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Leuprolide; Testosterone

INTERVENTIONS:
Drug: leuprolide
Drug: testosterone

SUMMARY:
OBJECTIVES:

I. Evaluate the effects of androgen suppression with leuprolide and androgen replacement with testosterone enanthate on muscle strength in men with Kennedy's disease or other motor neuron disease.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

All patients receive androgen suppression with leuprolide acetate injections every 4 weeks for 6 months, plus hormone replacement therapy with testosterone enanthate injections every week for 24 weeks.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Men aged 18 and over with motor neuron disease, i.e.:

* X-linked spinal and bulbar muscular atrophy (Kennedy's disease)
* Confirmed by androgen receptor, exon-1 mutation genotype
* Amyotrophic lateral sclerosis
* Spinal muscular atrophy

Significant muscle weakness on manual muscle testing

No prisoners

No mental disability

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 1992-10

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R. Mendell, Study Chair — Ohio State University